CLINICAL TRIAL: NCT05311371
Title: The Effect of Breathing Exercise on Chemotherapy-induced Nausea and Vomiting in With Autologous Hematopoietic Stem Cell Transplantation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Koc University Hospital (Other)
Responsible Party: Principal Investigator, ZELİHA GENÇ, Principal Investigator and PhD thesis student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022.065.IRB1.034
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Nausea; Vomiting; Breathing exercise; Autologous Hematopoietic Stem Cell Transplantation; Chemotherapy
MeSH Terms: conditions — Vomiting; Nausea | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: All of the participants were blinded to the randomization procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing exercise group (Experimental): The researcher will collect the data using Patient Information Form, Rhodes Index of Nausea, Vomiting and Retching Scale, Patient Diary for determining the number of nausea, vomiting, and retching episodes and the hours of breathing exercise of the patient, and Daily Nutritional Consumption Amount Form through face-to-face interview technique on the first day and for 14 days.
  During chemotherapy and stem cell transplantation, antiemetic treatment included in the treatment protocol will be applied to the patients.
  The patients will train about the application of breathing exercise by the researcher. They will be asked to do this breathing exercise with the guideline for at least 5 min in case of sensation of nausea and vomiting for 14 days.
  Interventions: Other: Breathing exercise group
- Control group (Other): The researcher will collect the data using Patient Information Form, Rhodes Index of Nausea, Vomiting and Retching Scale, Patient Diary for determining the number of nausea, vomiting, and retching episodes and the hours of breathing exercise of the patient, and Daily Nutritional Consumption Amount Form through face-to-face interview technique on the first day. The researcher will continue to fill out Rhodes Index of Nausea, Vomiting and Retching Scale, Patient Diary for determining the number of nausea, vomiting, and retching episodes and the hours of breathing exercise of the patient, and Daily Nutritional Consumption Amount Form for 14 days.
  During chemotherapy and stem cell transplantation, antiemetic treatment included in the treatment protocol will be applied to the patients.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Breathing exercise group — The exercise was applied in accordance with the "Guideline on Breathing Exercise for Reducing Nausea and Vomiting" prepared by the researcher in accordance with the literature. In addition, the researcher has a breath coaching certificate. The guideline include the application steps of breathing exercise. First, the researcher will demonstrate to the patients the practice of breathing exercise in accordance with the guideline. In the next step, patients they will be asked to do this application on themselves. The training is planned to take about 15-20 minutes for each patient. This guide will be given to patients after the training. They will be asked to do this breathing exercise correctly and effectively in accordance with the guideline for at least 5 min in case of sensation of nausea and vomiting for 14 days. The researcher will follow up the patients for 14 days by visiting room them every day.
  Arms: Breathing exercise group
Other: Control group — No intervention
  Arms: Control group

SUMMARY:
Nausea and vomiting are serious problems in patients undergoing autologous stem cell transplantation. It is stated that the incidence of acute and delayed nausea and vomiting is more than 50%, even if the patient has been given antiemetic prophylaxis during the treatment process.

Breathing is the easiest relaxation exercise applied during the flow in everyday life and also one of the most important and essential parts of other relaxation exercise. The handbooks prepared for the patients undergoing chemotherapy recommend deep breathing exercises in order to prevent their nausea and vomiting.

The aim of this study is to determine the effect of respiratory exercise on chemotherapy-induced nausea and vomiting in patients with autologous hematopoietic stem cell transplantation.

Research Hypotheses Ho: Respiratory exercise is not effective in preventing chemotherapy-associated nausea and vomiting in autologous hematopoietic stem cell transplant patients.

H1: Respiratory exercise is effective in preventing chemotherapy-associated nausea and vomiting in autologous hematopoietic stem cell transplant patients.

In the literature, no study has been found investigating the effect of breathing exercises on chemotherapy-induced nausea and vomiting for autologous hematopoietic stem cell transplantation patients.

The aim of this study is to determine the effect of respiratory exercise on chemotherapy-induced nausea and vomiting in patients with autologous hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Least 18-years-old,
* Autologous hematopoietic stem cell transplantation and take high-dose chemotherapy,
* not have any communicative problems,
* not have Coronavirus disease (COVID-19) disease or respiratory disease,
* Hb value of 10 and above and
* knowing how to read, write, and speak Turkish

Exclusion Criteria:

* have respiratory disease and Coronavirus disease (COVID-19),
* having any communication and psychiatric problem,
* not knowing how to read, write, and speak Turkish,
* not wanting to participate in the study and have anemia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — least 18-years-old
Enrollment: 70 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | Baseline
  Patient Information Form is a form prepared to determine the sociodemographic and disease-related characteristics of the patients. Sociodemographic characteristics of patient are composed of height, age, weight, educational status, social security, occupation, marital status, nutritional habits, smoking and alcohol use. Patient Information Form have general information about the patients such as diagnosis, duration, stage, and metastasis status of the disease, antiemetic drugs and treatment history. Disease history of cancer is , nausea-vomiting complaints before chemotherapy, the presence of any non-pharmacological method used to reduce nausea and vomiting induced by chemotherapy drugs.

SECONDARY OUTCOMES:
Rhodes Index of Nausea, Vomiting ve Retching | Baseline and 14 days
  Responses to each item are classified by using expressions appropriate to the item and scoring the severity of the nausea-vomiting-retching experience from 0 to 4. There are eight items in this scale that evaluate the experience, frequency and distress of nausea-vomiting and retching. The increase in score reflects worsening of the complaint experienced.

OTHER OUTCOMES:
Daily Nutritional Consumption Amount Form | Baseline and 14 days
  The amount of consumption of the patient in the morning, lunch, evening and snacks will be recorded before the treatment and throughout the study. The patient's antiemetic treatment, enteral and parenteral nutrition will be recorded daily in the follow-up form.
Patient Nausea And Vomiting Episode Follow-Up Form | Baseline and 14 days
  This follow-up chart was created by the researcher in order to evaluate the severity and episode of nausea and vomiting symptom during chemotherapy treatment and post-transplantation in patients with autologous hematopoietic stem cell transplantation. The scale consists of a 100 mm/10 cm long horizontal line. On the left end of the line, there is 0 "No nausea" statement, while on the right end there is 10 "Nausea is very severe" statement.
  The patient will be asked to mark the point on the line that will accurately reflect his or her nausea state. In addition, the patient will be asked to write down the number of nausea and vomiting numerically.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen L, de Moor CA, Eisenberg P, Ming EE, Hu H. Chemotherapy-induced nausea and vomiting: incidence and impact on patient quality of life at community oncology settings. Support Care Cancer. 2007 May;15(5):497-503. doi: 10.1007/s00520-006-0173-z. Epub 2006 Nov 14. PMID 17103197
- [Result] Haiderali A, Menditto L, Good M, Teitelbaum A, Wegner J. Impact on daily functioning and indirect/direct costs associated with chemotherapy-induced nausea and vomiting (CINV) in a U.S. population. Support Care Cancer. 2011 Jun;19(6):843-51. doi: 10.1007/s00520-010-0915-9. Epub 2010 Jun 9. PMID 20532923
- [Result] Roila F, Molassiotis A, Herrstedt J, Aapro M, Gralla RJ, Bruera E, Clark-Snow RA, Dupuis LL, Einhorn LH, Feyer P, Hesketh PJ, Jordan K, Olver I, Rapoport BL, Roscoe J, Ruhlmann CH, Walsh D, Warr D, van der Wetering M; participants of the MASCC/ESMO Consensus Conference Copenhagen 2015. 2016 MASCC and ESMO guideline update for the prevention of chemotherapy- and radiotherapy-induced nausea and vomiting and of nausea and vomiting in advanced cancer patients. Ann Oncol. 2016 Sep;27(suppl 5):v119-v133. doi: 10.1093/annonc/mdw270. No abstract available. PMID 27664248
- [Result] Rapoport BL. Delayed Chemotherapy-Induced Nausea and Vomiting: Pathogenesis, Incidence, and Current Management. Front Pharmacol. 2017 Jan 30;8:19. doi: 10.3389/fphar.2017.00019. eCollection 2017. PMID 28194109
- [Result] Aybar DO, Kilic SP, Cinkir HY. The effect of breathing exercise on nausea, vomiting and functional status in breast cancer patients undergoing chemotherapy. Complement Ther Clin Pract. 2020 Aug;40:101213. doi: 10.1016/j.ctcp.2020.101213. Epub 2020 Jun 14. PMID 32891289
- [Result] Suryono A., Akbar F., Nugraha F.S., Armiyati Y. Combination of of deep breathing relaxation and murottal reducing post chemotherapy nausea intensity in nasopharyngeal cancer (NPC) patients, Media Keperawatan Indonesia. 2020; 3: 24-31.
- [Result] Yoo HJ, Ahn SH, Kim SB, Kim WK, Han OS. Efficacy of progressive muscle relaxation training and guided imagery in reducing chemotherapy side effects in patients with breast cancer and in improving their quality of life. Support Care Cancer. 2005 Oct;13(10):826-33. doi: 10.1007/s00520-005-0806-7. Epub 2005 Apr 23. PMID 15856335